CLINICAL TRIAL: NCT00905736
Title: Influence of Microcurrent Parameters on Effectiveness of Treatment of Chronic Tennis Elbow - a Preliminary Trial
Brief Title: Influence of Microcurrent Parameters on Effectiveness in Treatment of Chronic Tennis Elbow
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Hertfordshire (Other)
Responsible Party: Leon Poltawski, University of Hertfordshire
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HEPEC/03/09/74
Record Dates: First submitted 2009-05-20; First posted 2009-05-21 (Estimated); Last update posted 2010-06-22 (Estimated); Status verified 2009-08

CONDITIONS: Tennis Elbow
Keywords: tendon; healing; microcurrent; chronic tennis elbow
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- current controlled (Experimental): a current controlled microcurent device providing a primarily monophasic waveform of typical amplitude 40 microamps
  Interventions: Procedure: Microcurrent treatment (controlled current)
- voltage controlled (Experimental): constant voltage amplitude delivering high frequency AC waveform
  Interventions: Procedure: Micocurrent treatment (controlled voltage)

INTERVENTIONS:
Procedure: Microcurrent treatment (controlled current) — primarily monophasic waveform of average amplitude 40 microamps, 1 hr daily for 3 weeks
  Arms: current controlled
Procedure: Micocurrent treatment (controlled voltage) — Microcurrent delivered for 6 hours daily for 3 weeks
  Arms: voltage controlled

SUMMARY:
Tennis elbow is a relatively common musculoskeletal disorder that can cause significant pain and disability. Treatment of the disorder is not always successful, and it often recurs or becomes chronic. More effective management options are required. There is evidence that electric microcurrent can promote tissue healing and symptom resolution in various chronic hard and soft tissue disorders, but few human studies have investigated its use with chronic tendon problems. It is an easily applied therapy with very few reports of side effects. It can be applied at home using a portable unit and, if it is clinically effective, may also prove more cost effective than other therapies.

A clinical trial is planned to evaluate the therapy but, in the absence of relevant published evidence, a preliminary study is required to look for a treatment effect and inform a power calculation for sample size, The study is comparing the effects of two different forms of microcurrent treatment.

ELIGIBILITY:
Inclusion Criteria:

* symptoms of tennis elbow for at least 3 months
* clinical diagnosis of tennis elbow

Exclusion Criteria:

* significant symptom improvement in previous month
* receipt of any active treatment for the condition in the previous month
* currently under the care of another health professional for tennis elbow
* current cervical radiculopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Tissue healing as indicated by sonography | baseline, 3 weeks, 6 weeks, 4 months

SECONDARY OUTCOMES:
Patient rating global change | baseline, 3 weeks, 6 weeks, 4 months
Pain free grip strength | baseline, 3 weeks, 6 weeks, 4 months
Patient rated tennis elbow questionnaire | baseline, 3 weeks, 6 weeks, 4 months
Adverse events | 3 weeks, 6 weeks, 4 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Hertfordshire, Hatfield, Hertfordshire, United Kingdom

REFERENCES:
- See also: application of electrotherapy — http://www.electrotherapy.org